CLINICAL TRIAL: NCT00549471
Title: Improvement After Botulinum Toxin A Injections to the Upper Extremities in Children With Cerebral Palsy
Brief Title: Improvement After Botulinum Toxin Injections to the Arms in Children With Cerebral Palsy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no funding
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Dr Van Dayk, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 180907.ctil
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Cerebral Palsy
Keywords: children with cerebral palsy ages eight to eleven.
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BG (Experimental): cooperative quadriplegic CP children ages 8-11 years, gross motor function level 4 with troublesome hypertonia that will respond to treatment. BG children will be given Botulinum Toxin A, as clinically required, in addition to an equivalent program of intensive therapy
  Interventions: Other: Botulinum Toxin A and physiotherapy
- Control Group (No Intervention): control group: Twenty cooperative quadriplegic CP children ages 8-11 years, gross motor function level 4 with troublesome hypertonia that will respond to treatment.CG children will undergo a program of intensive therapy.
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — CG children will undergo a program of intensive physiotherapy
  Arms: Control Group
Other: Botulinum Toxin A and physiotherapy — BG children will be given Botox, as clinically required, in addition to an equivalent program of intensive therapy. Botox injection will be tailored according to the specific child. Generally injection site will include biceps and brachioradialis, while flexors of the wrist and digits will be injected according to abnormal postures during function. Maximal total dose will be 23 IU per kg.
  Arms: BG

SUMMARY:
Hypothesis: (1) Treating upper limb hypertonia/spasticity with Botox®, in addition to reducing hypertonia/spasticity, will (a) improve global development, (b) improve function (passive & active), (c) reduce carer burden and (d) improve quality of life. (2) Early treatment with Botox® will have a greater impact on the rate of global development when compared to late treatment.

DETAILED DESCRIPTION:
Background: Upper limb function is essential for activities of daily living impacting on quality of life in children with cerebral palsy (CP). In preschool children, dysfunctional upper extremity manipulation not only leads to disability but may further delay global development and substantially increase career burden. Even modest functional improvement could have tremendous long-term benefit in activities of daily living and significantly reduce career burden. Hypertonia is the main symptom causing motor dysfunction in CP. Intramuscular Botulinum toxin injection is one way of treatment. In spite of anecdotal evidence suggesting that early intervention can lead to better outcomes, Israeli physicians are unable to prescribe this treatment for the upper extremities due to limited health insurance coverage. A paucity research evidence is often cited as the reason for limiting the insurance coverage, in particular to the upper limb. We therefore propose to study the effects of Botox® in treating children with CP.

Method: Twenty cooperative quadriplegic CP children ages 8-11 years, gross motor function level 4, will be enrolled for the study. Inclusion criteria will be troublesome hypertonia that will respond to treatment with Botox® (as identified by clinical assessment and neurophysiological measures). Since cooperation is crucial for the intensive therapy children with cognitive impairment (IQ<70) or severe behavioural disorders will be excluded. The children will be randomized to one of two groups a Botox group (BG) and a control group (CG). CG children will undergo a program of intensive therapy and BG children will be given Botox, as clinically required, in addition to an equivalent program of intensive therapy. Botox injection will be tailored according to the specific child. Generally injection site will include biceps and brachioradialis , while flexors of the wrist and digits will be injected according to abnormal postures during function. Maximal total dose will be 23 IU per kg. The intensive therapy will be as clinically required and the therapy program will be fully documented.

Outcome measures will include the following:

1. Hypertonia- neurophysiological measures
2. Impairment measures - Grip and Pinch strength, active and passive range of motion at the writs elbow and shoulder
3. Upper extremity function - Quality of Upper Extremity Skills Test (QUEST), Box and Blocks test
4. Function and patient needs assessment - Goal Attainment Scores, Developmental Fine Motor Scale, Pediatric Evaluation and Disability Inventory (PEDI)
5. Quality of life scales (care and comfort hypertonicity questionnaire) All of these measures will be taken once before treatment and then repeated at 7 months, and at 13 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* cooperative quadriplegic CP children
* gross motor function level 4
* troublesome hypertonia that will respond to treatment with Botox

Exclusion Criteria:

* cognitive impairment (IQ<70)
* severe behavioural disorder

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2007-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 2 years

SECONDARY OUTCOMES:
1. Hypertonia 2. Impairment measures 3. Upper extremity function 4. Function and patient needs assessment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hilla Ben-Pazi, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel